## Sublingual Estradiol Versus Oral Estradiol in Transgender Women

NCT04036500

Protocol last modified 3/14/2021

## **Sublingual Estradiol Versus Oral Estradiol in Transgender Women**

**Protocol Summary** 

Primary aim. To establish the pharmacokinetics of sublingual estradiol versus oral estradiol.

Secondary aim. To compare estradiol by LC-MS/MS to estradiol by immunoassay.

Design: To illuminate the pharmacokinetic parameters of sublingual estradiol in transgender women, a pilot crossover study will be conducted. Ten participants, transgender male-to-female patients who are naïve to hormone therapy, will be recruited from the Medical College of Wisconsin's Inclusion Health Clinic.

Methods: Each participant will be dosed with 1 mg oral estradiol. Blood will be drawn via a percutaneous intravenous catheter at hours 0,1,2,3,4,6,8. A wash-out period of at least one week will allow for complete clearance of the exogenous oral estradiol before testing the pharmacokinetics of sublingual estradiol 1 mg on the same ten patients in the same manner. Estradiol and estrone by LC-MS/MS will be measured, as well as estradiol by immunoassay. These will be sent to ARUP.